CLINICAL TRIAL: NCT01762475
Title: Sildenafil for the Treatment of Cerebrovascular Dysfunction During the Chronic Stage After Traumatic Brain Injury.
Brief Title: Sildenafil for Cerebrovascular Dysfunction in Chronic Traumatic Brain Injury.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Professor of Neurology, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T-N-2215; T-N-2215 (Other: NIH)
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Traumatic Brain Injury; Post-concussive Syndrome
Keywords: Magnetic resonance imaging; Blood oxygen level dependent signal; Hypercapnia; Endothelial progenitor cells
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome; Hypercapnia | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental: Group 1--Symptomatic TBI (Experimental): Experimental Group, Group 1, will consist of twenty-four male and female adult participants who have persistent TBI symptoms lasting more than six months.
  Participants in the experimental group will be randomized in a 1:1 ratio, assigned to group a or b.
  Participants randomized into Group 1a will take placebo twice daily for 8 weeks, followed by 8 weeks of sildenafil 25 mg twice daily with a 2-week washout period between the two 8-week periods.
  Participants randomized into Group 1b will take sildenafil 25 mg twice daily for 8 weeks, followed by 8 weeks of placebo twice daily with a 2-week washout period between the two treatment periods.
  Interventions: Drug: Sildenafil
- Active Comparator: Group 2--Healthy Controls (Active Comparator): Group 2 will be comprised of twenty male and female adult participants who have never experienced a TBI or concussion to serve as age and gender-matched healthy controls. Participants in Group 2 will have a single visit to measure cerebrovascular reactivity before and after a single dose of sildenafil (50 mg by mouth).
  Interventions: Drug: Sildenafil
- Group 3--Recovered TBI (Active Comparator): Group 3 will be comprised of twenty male and female adult participants who have experienced a TBI, have recovered, and are asymptomatic at the time of screening, to serve as age and gender-matched asymptomatic TBI controls. Participants in Group 3 will have a single visit to measure cerebrovascular reactivity before and after a single dose of sildenafil (50 mg by mouth).
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil
  Other Names: Viagra

SUMMARY:
The purpose of this study is to determine whether sildenafil (Viagra®) is effective in improving cerebral blood flow and cerebrovascular reactivity inpatients who have persistent symptoms at least 6 months after a traumatic brain injury (TBI).

DETAILED DESCRIPTION:
The goal of this Phase II study is to generate pilot data that will allow for the design of a clinical trial of sildenafil (Viagra®) to treat patients with traumatic vascular injury in the chronic state after traumatic brain injury (TBI). Injury to small and medium-sized blood cerebral blood vessels is a well-recognized consequence of traumatic brain injury (TBI). Non-invasive imaging with positron emission tomography (PET) and single photon emission computerized tomography (SPECT) have long demonstrated deficits in cerebral blood flow in TBI, including in symptomatic patients years after mild TBI (mTBI). Recently, magnetic resonance imaging (MRI) methods have been developed which allow reliable and non-invasive measurement of cerebrovascular reactivity (CVR) to vasodilatory stimuli such as hypercapnia in humans. These techniques have never been applied to symptomatic patients in the chronic stage after mTBI. These methods are particularly promising due to the recent discovery that phosphodiesterase-5 (PDE5) inhibitors improve cerebral blood flow, induce angiogenesis and neurogenesis, and improve functional recovery in animals after experimental stroke and cryoinjury. This pilot study will use novel MRI methods (Blood Oxygen Level Dependent (BOLD) response to hypercapnia) to noninvasively measure cerebrovascular reactivity in the chronic stage after TBI, and the first to use sildenafil in patients with chronic TBI.

The study has one primary objective and 10 secondary objectives:

Primary objective:

1. Single dose treatment with sildenafil (50 mg orally) is effective in increasing the global BOLD response to hypercapnia in symptomatic patients in the chronic stage after TBI.

   Secondary objective (Safety and Tolerability):
2. Sildenafil therapy (25 mg orally twice daily) is well tolerated in symptomatic patients in the chronic stage after TBI, with few adverse effects and treatment discontinuations in less than 10% of patients.

   Tertiary (Exploratory) objectives:
3. Single dose treatment with sildenafil (50 mg orally) is effective in increasing the regional BOLD response to hypercapnia in symptomatic patients in the chronic stage after TBI.
4. Patients with persistent symptoms in the chronic stage after TBI have deficits in cerebrovascular reactivity compared to uninjured healthy controls.
5. Patients with persistent symptoms in the chronic stage after TBI have deficits in cerebrovascular reactivity compared to asymptomatic patients after TBI.
6. Patients with persistent symptoms in the chronic stage after TBI have reduced numbers of circulating EPCs compared to uninjured healthy controls.
7. Patients with persistent symptoms in the chronic stage after TBI have reduced numbers of circulating EPCs compared to asymptomatic patients after TBI.
8. The effect on cerebrovascular reactivity of single dose treatment with sildenafil persists after 8 weeks of chronic therapy (25 mg orally, twice daily).
9. Treatment with sildenafil for 8 weeks (25 mg orally twice daily) increases the number of circulating endothelial progenitor cells (EPCs) in symptomatic chronic TBI patients.
10. Treatment with sildenafil for 8 weeks (25 mg orally twice daily) reduces the prevalence of post-concussive symptoms, compared to placebo treatment.
11. Treatment with sildenafil for 8 weeks (25 mg orally twice daily) improves performance in neuropsychometric tests, compared to placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria applied to all participants

In order to be included in this study, all participants must meet the following minimum criteria:

1. Age 18 - 55 years, inclusive
2. Ability to undergo MRI scanning.
3. Ability to read, write, and speak English.
4. Stable doses of concomitant medications for at least 2 weeks prior to enrollment.
5. Likelihood of completing 18 weeks of study procedures. Likelihood of ability to complete the study procedures means that the person has 1) a low probability of being deployed during the 18-week period 2) verbalizes intent to complete the study.

Inclusion Criteria for Group 1 (symptomatic TBI)

In order to be included in the symptomatic TBI Group, study participants must meet the following criteria:

1. A history of having sustained a TBI > 6 months and < 10 years prior to enrollment. Evidence will be any one of the following 3 criteria:

   1. GCS 3 - 12 (GCS obtained in Emergency Room and noted in medical record)
   2. Post-traumatic amnesia > 24 hours
   3. TBI-related abnormality on neuroimaging (either CT or MRI). (Some missing information about the initial injury (i.e. documentation of initial GCS) is not necessarily exclusionary if the bulk of the available history is indicative that the patient suffered a TBI and meets the inclusion criteria)
2. Persistent post-concussive symptoms, according to the DSM-IV Research Criteria for Post-Concussional Disorder, including:

   1. Evidence from neuropsychological testing of difficulty in attention or memory. (refers to neuropsychological testing done as a part of the patient's hospital or rehabilitation care not as a part of screening for this study)
   2. Three or more of the following symptoms, which started shortly after the trauma and persist for at least three months:

   i) Fatigability ii) Disordered sleep iii) Headache iv) Vertigo or dizziness v) Irritability or aggression vi) Anxiety, depression, or affective instability vii) Changes in personality (e.g. social or sexual inappropriateness) viii) Apathy or lack of spontaneity c) Symptoms in criteria (a) and (b) must have their onset after trauma, or there was a significant worsening of pre-existing symptoms after trauma.

   d) Disturbance from these symptoms causes significant impairment of social or occupational functioning and represents a significant decline from previous level of functioning.

   Inclusion Criteria Group 2-Healthy controls In order to be included in this study, participants must meet the inclusion criteria for all participants listed in 4.2.

   3.2.3 Inclusion Criteria Group 3-Recovered TBI

1. History of having sustained a TBI > 6 months and < 10 years prior to enrollment. This evidence will be any one of the following:

a) GCS 3 - 12 (GCS obtained in Emergency Room after injury and noted in medical record) b) Post-traumatic amnesia > 24 hours c) TBI-related abnormality on neuroimaging (either CT or MRI) 2. Does not meet criteria for persistent post-concussive symptoms, according to the DSM-IV Research Criteria for Post-concussional Disorder defined by the following:

1. No evidence from neuropsychological testing of difficulty in attention or memory.
2. No more than 1 of the following symptoms, which started shortly after the trauma and persists for at least three months:

i) Fatigability ii) Disordered sleep iii) Headache iv) Vertigo or dizziness v) Irritability or aggression vi) Anxiety, depression, or affective instability vii) Changes in personality (e.g. social or sexual inappropriateness) viii) Apathy or lack of spontaneity c) No impairment of social or occupational functioning or a significant decline from previous level of functioning.

Exclusion Criteria:

Exclusion Criteria for all Groups:

1. Contraindication to sildenafil which includes the following:

   1. Current use of organic nitrate vasodilators
   2. use of ritonavir (HIV-protease inhibitor)
   3. Current use of erythromycin, ketoconazole, or itraconazole
   4. Current use of cimetidine
   5. Alpha-blockers such as doxazosin (Cardura), tamsulosin (Flomax), and terazosin (Hytrin) prazosin (Minipres). These medications are usually used for the treatment of enlarged prostate.
   6. Current resting hypotension (BP < 90/50 mm Hg)
   7. Current severe renal insufficiency (Creatinine Clearance < 30 mL/min)
   8. Current hepatic cirrhosis
   9. Current cardiac failure or coronary artery disease causing unstable angina
   10. Retinitis pigmentosa
   11. Known hypersensitivity or allergy to sildenafil or any component of the tablet
2. Evidence of penetrating injury
3. Daily therapy with a PDE5 inhibitor within the past 2 months
4. History or evidence of pre-existing neurological or psychiatric disorder not related to TBI, such as:

   1. Multiple sclerosis, pre- or co-existing
   2. Stroke (other than stroke at the time of TBI)
   3. Pre-existing developmental disorder
   4. Pre-existing epilepsy
   5. Pre-existing major depressive disorder
   6. Pre-existing schizophrenia
5. Women who are pregnant or breast-feeding.

Exclusion for Healthy Control Group Any evidence or history of a TBI or concussion is exclusionary for the Control Group.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular reactivity | 24 months
  Single dose treatment with sildenafil (50 mg orally) is effective in increasing the global BOLD response to hypercapnia in symptomatic patients in the chronic stage after TBI.

SECONDARY OUTCOMES:
Safety and tolerability | 24 months
  Sildenafil therapy (25 mg orally twice daily) is well tolerated in symptomatic patients in the chronic stage after TBI, with few adverse effects and treatment discontinuations in less than 10% of patients.

OTHER OUTCOMES:
Regional cerebrovascular reactivity | 24 months
  Single dose treatment with sildenafil (50 mg orally) is effective in increasing the regional BOLD response to hypercapnia in symptomatic patients in the chronic stage after TBI.
Cerebrovascular reactivity in TBI patients vs. healthy controls | 24 months
  Patients with persistent symptoms in the chronic stage after TBI have deficits in cerebrovascular reactivity compared to uninjured healthy controls.
Cerebrovascular reactivity in symptomatic TBI vs. asymptomatic TBI | 24 months
  Patients with persistent symptoms in the chronic stage after TBI have deficits in cerebrovascular reactivity compared to asymptomatic patients after TBI.
Endothelial progenitor cells in TBI vs. healthy controls | 24 months
  Patients with persistent symptoms in the chronic stage after TBI have reduced numbers of circulating EPCs compared to uninjured healthy controls.
Endothelial progenitor cells in symptomatic TBI vs. asymptomatic TBI | 24 months
  Patients with persistent symptoms in the chronic stage after TBI have reduced numbers of circulating EPCs compared to asymptomatic patients after TBI.
Persistence of cerebrovascular reactivity effect. | 24 months
  The effect on cerebrovascular reactivity of single dose treatment with sildenafil persists after 8 weeks of chronic therapy (25 mg orally, twice daily).
Persistence of endothelial progenitor cell effect. | 24 months
  Treatment with sildenafil for 8 weeks (25 mg orally twice daily) increases the number of circulating endothelial progenitor cells (EPCs) in symptomatic chronic TBI patients.
Benefit on post-concussive symptoms | 24 months
  Treatment with sildenafil for 8 weeks (25 mg orally twice daily) reduces the prevalence of post-concussive symptoms, compared to placebo treatment.
Benefit on neuropsychologic testing | 24 months
  Treatment with sildenafil for 8 weeks (25 mg orally twice daily) improves performance in neuropsychometric tests, compared to placebo treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon R. Diaz-Arrastia, MD, PhD, Study Director — Uniformed Services University of the Health Sciences; Eric Wassermann, MD, Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institute of Health, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Reddy P, Izzetoglu M, Shewokis PA, Sangobowale M, Diaz-Arrastia R, Izzetoglu K. Evaluation of fNIRS signal components elicited by cognitive and hypercapnic stimuli. Sci Rep. 2021 Dec 6;11(1):23457. doi: 10.1038/s41598-021-02076-7. PMID 34873185